CLINICAL TRIAL: NCT01975935
Title: Clinical Protocol to Investigate the Efficacy of Amlexanox vs. Placebo for Treatment of Glucose and Lipid Abnormalities in Obese Type 2 Diabetics
Brief Title: Efficacy of Amlexanox vs. Placebo in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Elif Oral, Associate Professor, Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00079381
Record Dates: First submitted 2013-10-29; First posted 2013-11-05 (Estimated); Results first posted 2017-05-09 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus Type 2; Non-alcoholic Fatty Liver Disease; Obesity
Keywords: diabetes mellitus type 2; non-alcoholic fatt liver disease; obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease; Obesity | interventions — amlexanox

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablet (TID) 2 weeks Placebo tablets (2 x TID) 10 weeks
  Interventions: Drug: Placebo
- Amlexanox (Experimental): Solfa tablets (Amlexanox 25mg) TID for 2 weeks Solfa tablets (Amlexanox 25mg x 2) TID for 10 weeks
  Interventions: Drug: Amlexanox

INTERVENTIONS:
Drug: Amlexanox — 25 mg amlexanox tablets blinded by encapsulation
  Other Names: Solfa tablets
  Arms: Amlexanox
Drug: Placebo — placebo sham blinded by encapsulation in the same capsules as the study drug arm
  Arms: Placebo

SUMMARY:
This study involves research about an investigational medicine called Amlexanox. The reason for this study is to find out how Amlexanox can improve type 2 diabetes, insulin resistance, obesity and non-alcoholic fatty liver disease (NAFLD). In this study, Amlexanox is considered to be investigational (not approved by the Food and Drug Administration [FDA]) for type 2 diabetes, insulin resistance, obesity and non-alcoholic fatty liver disease (NAFLD). This is a placebo controlled study. There is a 50-50 chance that the patient may either receive the study drug, Amlexanox, or a placebo (sugar pill). Neither the patient or the study doctors will know if the patient is receiving the study drug or placebo.

DETAILED DESCRIPTION:
This proposal focuses on a clinical proof of concept study to evaluate a novel hypothesis. We propose that overnutrition, leading to obesity, represents a state of excessive energy storage promoted by insulin. The stress of excessive energy storage initiates a set of homeostatic responses that includes the generation of adipose tissue and liver inflammation, which involves the secretion of proinflammatory cytokines that block energy storage in fat and liver by inducing insulin resistance, thus relieving stress on the adipocyte and hepatocyte. However, our recent data suggest that inflammation itself is countered by a secondary feedback loop, which we have termed "counter-inflammation". We propose that this process keeps inflammation in check, ensuring that it is maintained at low levels. At the same time counter-inflammation also promotes energy conservation via increased energy storage and decreased utilization in a manner that is insulin-independent. We hypothesize that the noncanonical IkB kinases Ikke and TBK1 are "counterinflammatory" kinases that feedback inhibit inflammatory pathways while helping to support a positive energy balance.

How can this hypothesis be addressed in human subjects? A number of clinical trials have already been initiated with the intention of improving insulin resistance by attenuating inflammation. Many of these have focused on the blockade of single cytokines or their receptors such as TNFa, IL1 and MCP1 (CCR2 antagonist). While the record on these trials is mixed, the complexity of inflammatory pathways elicited during obesity suggests that inhibition of only a single cytokine is not likely to be sufficient. Additionally, because numerous studies have implicated the NFkB pathway in obesity-induced inflammation, NFkB inhibitors have been contemplated. Salsalate was originally resuscitated due to its perceived activity to block NFkB and hence to block inflammation. However, although clinical studies on this drug have been promising, precisely how salsalate works, what its target is, and whether it actually functions an NFkB inhibitor remains controversial (recent data indicate that it may act via activation of AMPK).

We describe here a new potential therapeutic agent that is the result of an academic collaborative drug discovery effort carried out at the University of Michigan. Our studies on elucidating the role of NFkB in insulin resistance and macrophage activation led to the identification of Ikke and TBK1 as potential targets for therapeutic intervention in obesity and type 2 diabetes. We performed a high throughput screen searching for inhibitors of these kinases, evaluating a group of 175,000 compounds that included a collection of approved drugs. Interestingly, the most potent and specific inhibitor discovered was amlexanox; an older drug originally developed in Japan for the treatment of asthma and allergic rhinitis, and later in the US for aphthous ulcers, but without a well understood mechanism of action. It has been in use since 1987, and has a favorable side effect profile.

This protocol is the first proof of concept study to evaluate the possible repurposing of Amlexanox for the treatment of type 2 diabetes and obesity. At the same time, we hope to test the hypothesis that IKKe and TBK1 may be important players in maintaining a positive energy balance, and also in supporting insulin resistance, during prolonged over-nutrition. Finally, these studies will also provide valuable insight into the validity of these two protein kinases as drug targets for the future development of new chemical entities useful in the treatment of type 2 diabetes. Therefore our specific aims are

1. Does amlexanox treatment improve measures of type 2 diabetes, insulin resistance and obesity? To address this question, we intend to treat patients with clinical Type 2 diabetes and Grade 1/2 obesity (BMI 27 to 45 kg/m2) for a period of 3 months in a double-blinded placebo controlled proof-of concept study. We will enroll 40 patients without evidence of severe end-organ damage from chronic complications of Type 2 diabetes who also are on metformin and/or DPPIV inhibitors or no medications, who also have clear-cut evidence of hyperglycemia (HbA1c>6.5% and <10.0%). These patients will be treated with either placebo or Amlexanox oral tablets at a starting dose of 25 mg PO tid for 2 weeks and then titrated up to a dose of 50 mg PO tid (doses used to treat asthma in humans and leading to serum concentrations comparable to metabolically effective doses in rodent studies) for the remainder of the therapy period. HbA1c is targeted as primary end-point in this study. Fasting lipid profiles, plasma insulin, HOMA-IR, clinical markers of inflammation and adipocytokine profiles will be measured as other parameters of interest at baseline, 6 weeks and 12 weeks. Insulin secretion as well as insulin sensitivity will be probed using a mixed meal test. Weight is also an important but secondary end-point in this study. We will determine resting energy expenditure with indirect calorimetry and total body composition using DEXA at baseline and 12 weeks. Safety monitoring with CBC, comprehensive metabolic biochemistry, CPK and urine analyses will be undertaken at 1, 2, 4, 6, and 12 weeks, and urinary albumin at baseline and 12 weeks. Measures of safety and efficacy will be repeated 4 weeks after the drug has been discontinued as well.
2. Does amlexanox treatment improve measures of NAFLD in obese patients? All participants in the clinical proof-of-concept study outlined in the aim above will be studied for the degree of steatosis in the liver with the use of MRI and MR spectroscopy at baseline and at 3 months of the study.
3. Development of biomarkers for treatment of patients with type 2 diabetes by amlexanox. We will evaluate the phosphorylation of proteins known to be targets of IKKe and TBK1 in blood, and adipose tissue samples. We will use phospho-specific antibodies to evaluate the regulation of targets that play a role in energy metabolism, and also in feedback inhibition of NFkB. These studies will pave the way for future evaluations probing the metabolic relevance of IKKe and TBK1 in humans using the same agent or more potent ones to be discovered or designed.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old at baseline.
* Is male, female not of childbearing potential, or meets all the following criteria if female of childbearing potential (including perimenopausal women who have had a menstrual period within one year):

  * Not breastfeeding.
  * Negative pregnancy test result (human chorionic gonadotropin, beta subunit [βhCG]) at baseline (not applicable to hysterectomized females).
  * Must practice and be willing to continue to practice appropriate birth control (defined as a method which results in a low failure rate when use consistently and correctly, such as implants, injectables, oral contraceptives, some intrauterine contraceptive devices, sexual abstinence, tubal ligation, or a vasectomized partner) during the entire duration of study period.
* Has physician-confirmed diabetes mellitus with a clear diagnosis or per ADA criteria with fasting glucose>126 mg/dL or HbA1c >6.4% or 2 hour GTT >200 mg/dL.
* BMI ≥27 and <45 kg/m2.
* On no medications or only on first line oral medications (such as Metformin and/or DPP IV inhibitors) for treatment of Type 2 diabetes mellitus with a stable regimen for >12 weeks.
* Alcohol consumption of less than 40 grams/week.
* A liver US confirming presence of fatty infiltration of the liver.
* Is able to read, understand and sign the U of M IRBMED approved informed consent form (ICF), communicate with study physician and study team, understand and comply with protocol requirements.

Exclusion Criteria:

* On insulin, or other injectables for treatment of Type 2 diabetes.
* Unable to conduct home based glucose monitoring.
* HbA1c <6.5% and >10.0% (set to achieve uniformity in the study population).
* Presence of advanced liver disease (as evidenced by abnormal synthetic function, abnormal PT or albumin).
* Evidence of other etiologies of viral hepatitis.
* Presence of hematologic, bone marrow and/or other abnormalities.
* Presence of hemoglobinopathy or other hematological abnormalities that will interfere with accurate measurement of HbA1c.
* Presence of HIV infection.
* Inability to give informed consent.
* Presence of ESRD, any type of active cancer, or >class 2 congestive heart failure ((New York Heart Association Functional Classification System), based on medical history and physical examination.
* Active chronic infection such as known chronic osteomyelitis or tb, etc. (may be transient).
* Creatinine >1.5 mg/dL.
* Proliferative diabetic retinopathy, nonproliferative retinopathy is allowed.
* Unable to ambulate.
* Clinically relevant CAD: history of stent, CABG or cardiologist confirmed angina.
* Any other condition in the opinion of the investigators that may impede successful data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-01; Primary Completion 2016-04-25 (Actual); Study Completion 2017-08-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo tablet (TID) 2 weeks Placebo tablets (2 x TID) 10 weeks
  Placebo
- Amlexanox: Solfa tablets (Amlexanox 25mg) TID for 2 weeks Solfa tablets (Amlexanox 25mg x 2) TID for 10 weeks
  Amlexanox
Period: Overall Study
Arm/Group | Placebo | Amlexanox
Started | 21 | 21
Completed | 18 | 20
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Amlexanox | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 18 | 35
  >=65 years | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.24 (7.65) | 55.81 (9.52) | 57.52 (8.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 11 | 11 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 19 | 19 | 38
  African American | 2 | 1 | 3
  Asian | 0 | 1 | 1
  Native American | 0 | 0 | 0
  Unknown | 0 | 0 | 0
  Decline to Answer | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Difference in Hemoglobin A1c Values
Description: Difference in hemoglobin A1c as measured at baseline and week 12 visits
Time Frame: 12 weeks (measured at baseline and 12 weeks)
Population: The number of participants analyzed at week 12 differs from the overall number analyzed at baseline because 1 treatment group and 3 placebo group participants dropped from the study before their week 12 visit.
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin glycated
Arm/Group | Placebo | Amlexanox
Number analyzed (Participants) | 21 | 21
percentage of hemoglobin glycated
  Baseline | 7.77 (1.07) | 7.68 (0.97)
  Week 12: number analyzed (Participants) | 18 | 20
  Week 12 | 7.76 (1.23) | 7.44 (0.95)
Statistical Analysis 1: Comparison: Placebo vs Amlexanox; Test type: Superiority; p = 0.05, t-test, 2 sided — This is the calculated p value and not the threshold for statistical significance

2. Secondary Outcome: Hepatic Steatosis as Measured by MRI
Description: Improvement in hepatic steatosis by MRI is shown by a decrease in percent fat from baseline to week 12 visit.
Time Frame: 12 weeks
Population: One placebo patient was an early termination and did not have an MRI scan done at the 12 week visit. A total of 20 patients received MRI scans due to funding limitations.
Measure: Mean (Standard Deviation); unit: % fat
Arm/Group | Placebo | Amlexanox
Number analyzed (Participants) | 9 | 11
% fat
  Baseline | 12.82 (7.82) | 18 (9.67)
  Week 12: number analyzed (Participants) | 8 | 11
  Week 12 | 12.88 (8.66) | 16.22 (9.86)
Statistical Analysis 1: Comparison: Placebo vs Amlexanox; Test type: Superiority; p = 0.38, t-test, 2 sided

3. Secondary Outcome: Change in Weight
Description: Change in weight (kilograms) as measured at baseline and week 12 visits.
Time Frame: 12 week
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Placebo | Amlexanox
Number analyzed (Participants) | 21 | 21
kilograms
  Baseline | 100.24 (19.77) | 100.95 (15.18)
  Week 12: number analyzed (Participants) | 18 | 20
  Week 12 | 97.94 (18.83) | 100.81 (14.03)
Statistical Analysis 1: Comparison: Placebo vs Amlexanox; Test type: Superiority; p = 0.51, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: March 31, 2014-May 25, 2017. 2 years, 2 months
Arm/Group | Placebo | Amlexanox
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/21 | 1/21
Other Adverse Events (participants affected / at risk) | 16/21 | 15/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=21) | Amlexanox (N=21)
NSTEMI (Cardiac disorders) | 1 (1) | 0 (0)
Injured left leg playing football (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=21) | Amlexanox (N=21)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (2)
Head cold (Immune system disorders) | 4 (4) | 0 (0)
Skin rash (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (5)
Indigestion (Gastrointestinal disorders) | 2 (2) | 0 (0)
Worsening neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 5 (5) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Ankle edema (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 2 (2)
Elevated CK (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Itchy skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Optimal drug dose is yet to be defined. The dose and the treatment duration may not have been sufficient to reveal all the positive as well as negative effects of the drug. Effects of combination with other anti-diabetics is also unknown.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No